CLINICAL TRIAL: NCT02334813
Title: A Randomized Trial of Daily Prednisone Versus Pulsed Dexamethasone in Treatment-naïve Adult Patients With Immune Thrombocytopenia
Brief Title: Daily Prednisone Versus Pulsed Dexamethasone in Treatment-naïve Adult Patients With Immune Thrombocytopenia
Acronym: EIS2002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Ulrich Duehrsen, Univ.-Prof. Dr. med., University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIS2002
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: daily prednisone (Active Comparator): During the first week of treatment patients in both arms receive prednisone at 1 mg/kg/d. In arm A prednisone is continued at 1 mg/kg/d for a second week. If platelets increase to ≥50/nl, its dose is reduced to <25 mg/d by week 14 and <7.5 mg/d by week 20 according to a step-wise reduction scheme provided in the protocol. In patients without response after 2 weeks of treatment, the prednisone dose is increased to 2 mg/kg/d for another 2 weeks, then tapered as described above.
  Interventions: Drug: Prednisone
- Arm B: pulsed dexamethasone (Active Comparator): During the first week of treatment patients in both arms receive prednisone at 1 mg/kg/d. In arm B patients subsequently receive six 21-day courses of pulsed dexamethasone (0.6 mg/kg/d, days 1-4).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Prednisone — Continuous daily therapy
  Arms: Arm A: daily prednisone
Drug: Dexamethasone — 4-day pulses every 3 weeks
  Arms: Arm B: pulsed dexamethasone

SUMMARY:
Patients above age 18 with a first episode of immune thrombocytopenia are randomized 1:1 between 2-4 weeks of daily prednisone (1 mg/kg/d) with subsequent dose tapering (arm A) and six 3-week cycles of pulsed dexamethasone (0.6 mg/kg/d, days 1-4; arm B). The primary endpoint is duration of remission defined as platelets ≥50/nl.

DETAILED DESCRIPTION:
Patients above the age of 18 years with a first episode of immune thrombocytopenia (ITP) are eligible for inclusion, except pregnant women and patients unable to tolerate glucocorticoids. Diagnosis is made and treatment requirement defined according to the 1996 practice guidelines of the American Society of Hematology. The primary endpoint is duration of remission defined as platelets ≥50/nl. Secondary endpoints are response rate, complete remission (platelets ≥150/nl), cumulative cortisol equivalent dose (potency of prednisone / dexamethasone relative to cortisol: x 4 / x 30) and adverse events. During the first week of treatment all patients receive prednisone at 1 mg/kg/d. This period is used to confirm the diagnosis and identify patients with ITP secondary to lymphoproliferative, autoimmune (systemic lupus erythematosus, antiphospholipid syndrome) or infectious diseases (human immunodeficiency, hepatitis C, cytomegalovirus infection). Patients are stratified by age (cut-off: 50 years), gender and primary versus secondary ITP and then randomized 1:1 between daily prednisone (arm A) and pulsed dexamethasone (arm B). In arm A prednisone is continued at 1 mg/kg/d for a second week. If platelets increase to ≥50/nl, its dose is reduced to <25 mg/d by week 14 and <7.5 mg/d by week 20 according to a step-wise reduction scheme provided in the protocol. In patients without response after 2 weeks of treatment, the prednisone dose is increased to 2 mg/kg/d for another 2 weeks, then tapered as described above. In arm B patients receive six 21-day courses of pulsed dexamethasone (0.6 mg/kg/d, days 1-4). Patients failing to achieve or maintain a remission are switched to the alternative treatment arm (A: no response after 4 weeks of prednisone at 1-2 mg/kg/d, loss of response, maintenance doses exceeding the above limits; B: no response after 2 cycles, loss of response).

ELIGIBILITY:
Inclusion Criteria:

* First episode of ITP

Exclusion Criteria:

* Pregnancy
* Glucocorticoid intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Dührsen, MD, Principal Investigator — University Hospital, Essen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Daily Prednisone | Arm B: Pulsed Dexamethasone
Started | 12 | 14
Completed | 9 | 13
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Daily Prednisone | Arm B: Pulsed Dexamethasone | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Median (Full Range); unit: years] | 43 [29 to 65] | 46 [22 to 77] | 44 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Remission Duration
Description: Percentage of patients in ongoing remission at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Daily Prednisone | Arm B: Pulsed Dexamethasone
Number analyzed (Participants) | 9 | 13
Participants | 3 | 11

ADVERSE EVENTS:
Arm/Group | Arm A: Daily Prednisone | Arm B: Pulsed Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 2/9 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Daily Prednisone (N=9) | Arm B: Pulsed Dexamethasone (N=13)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes